CLINICAL TRIAL: NCT05942456
Title: An Exploratory Research of Soluble B7-H3 Expression in Peripheral Blood as a Biomarker to Monitor Therapeutic Effect of Systemic Treatment for Osteosarcoma
Brief Title: Soluble B7-H3 as a Biomarker for Osteosarcoma
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Musculoskeletal Tumor Center, Peking University People's Hospital
Other Study IDs: PKUPH-sarcoma 16
Record Dates: First submitted 2023-07-05; First posted 2023-07-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Biomarker; Progression; Osteosarcoma; Surveillance
Keywords: sB7-H3; osteosarcoma; biomarker; prognosis; clinical evaluation
MeSH Terms: conditions — Disease Progression; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sB7-H3 of treatment-naive osteosarcoma patients: Before delivering neoadjuvant chemotherapy, using ELISA to test the protein expression of sB7-H3 of Peripheral Blood
  Interventions: Diagnostic Test: ELISA: enzyme-linked immunosorbent assay
- sB7-H3 after neoadjuvant chemotherapy for osteosarcoma patients: After neoadjuvant chemotherapy and before definitive surgery, using ELISA to test the protein expression of sB7-H3 of Peripheral Blood
  Interventions: Diagnostic Test: ELISA: enzyme-linked immunosorbent assay

INTERVENTIONS:
Diagnostic Test: ELISA: enzyme-linked immunosorbent assay — enzyme-linked immunosorbent assay

SUMMARY:
Increasing data has indicated an association between increased soluble B7-H3 (sB7-H3) levels and unfavorable prognosis in patients with malignancies. However, the level of sB7-H3 and its clinical significance in osteosarcoma are not well known. In this present study, we investigated whether sB7-H3 levels in serum could be as a biomarker for osteosarcoma treatment.

ELIGIBILITY:
Inclusion Criteria:

* High Grade osteosarcoma verified with pathologic diagnosis.
* systemic treatment-naive before the first time Blood drawing.
* ECOG 0 or 1 and all the other imagings indicate that patients could tolerate standard PKUPH-OS-02 protocol neoadjuvant chemotherapy.
* All radiographs are complete for clinical evaluation.

Exclusion Criteria:

* Patients who Can't tolerate blood drawing.
* Patients without complete medical records in PKUPH system.
* Patients who can't tolerate PKUPH-OS-02 neoadjuvant chemotherapy.
* other conditions that investigators think are not suitable for this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initial treated osteosarcoma patients in PKUPH and later would recieve definitive surgery in PKUPH with complete clinical materials.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation of quantity of Protein B7-H3 Expression with clinical evaluation | 6 months
  Clinical evaluation according to RECIST 1.1

SECONDARY OUTCOMES:
correlation of quantity of Protein B7-H3 Expression with histological responses | 6 months
  Histological responses according to Huvos Grade
correlation of quantity of Protein B7-H3 Expression with event-free survival | 2 years
  event-free survival calculated from starting systemic therapy to any tumor-related events for progression
correlation of quantity of Protein B7-H3 Expression with overall survival | 5 years
  overall survival calculated from starting systemic therapy to death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang L, Kang FB, Zhang GC, Wang J, Xie MF, Zhang YZ. Clinical significance of serum soluble B7-H3 in patients with osteosarcoma. Cancer Cell Int. 2018 Aug 13;18:115. doi: 10.1186/s12935-018-0614-z. eCollection 2018. PMID 30123093
- [Background] Xie L, Chen C, Liang X, Xu J, Sun X, Sun K, Yang R, Tang X, Guo W. Expression and Clinical Significance of Various Checkpoint Molecules in Advanced Osteosarcoma: Possibilities for Novel Immunotherapy. Orthop Surg. 2023 Mar;15(3):829-838. doi: 10.1111/os.13620. Epub 2022 Dec 15. PMID 36519392